CLINICAL TRIAL: NCT03045588
Title: The Effects of a Train High, Sleep Low Strategy on Performance, Substrate Utilization and Muscular Adaptations in Moderately Trained Cyclists
Brief Title: The Effects of a Train High, Sleep Low Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Team Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sleep low
Record Dates: First submitted 2017-01-29; First posted 2017-02-07 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Cycling Performance; Muscular Adaptations; Substrate Utilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low group (Experimental): This subjects in this group conducts all their morning exercise sessions with high fat oxidation (in a fasted condition). Thus, the subjects in this group after high intensity exercise in the evening do not get any carbohydrates to eat after training until the exercise session the following morning has been conducted.
  Interventions: Other: Combined exercise and diet intervention
- High group (Active Comparator): This subjects in this group conducts all their morning exercise sessions with low fat oxidation (in a fed condition). Thus, the subjects in this group after high intensity exercise in the evening do get carbohydrates to eat after training until the exercise session the following morning has been conducted.
  Interventions: Other: Combined exercise and diet intervention

INTERVENTIONS:
Other: Combined exercise and diet intervention — Both groups exercise 6 times per week in 4 weeks conducted as 3 evening and 3 morning sessions per week. Both groups receive dietary products to be consumed immediately before and after each evening and morning session, respectively. One group conduct morning sessions in a fasted state, the other conduct the morning sessions in a fed state. Performance pre and post is measured, and muscle biopsies are obtained.

SUMMARY:
The investigators will examine the long-term effects of a combined training and diet intervention that, acutely, increases fat oxidation during exercise. This is done with a 4 week intervention study with moderately trained cyclists. Performance is tested pre and post intervention and muscle biopsies are obtained.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* VO2-max>55 ml/kg/min
* No smokers
* Training 6 hours per week (cycling)
* Training experience for more than 3 years.

Exclusion Criteria:

* Less than 2 g carbohydrate/kg/day

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Time trial performance measured in Watts | Change from Baseline and after 4 weeks of training
  30 min time trial after 90 minutes of intensive cycling. The average amount of Watts during the 30 minutes will be measured.

SECONDARY OUTCOMES:
Protein expression in skeletal muscle tissue | Baseline and after 4 weeks of training
  Amount of mitochondrial proteins and enzymes will be measured with a Western Blotting technique
The absolute amount of carbohydrate and fat which is metabolised during morning exercise, measured in grams/minute | Baseline and after 4 weeks of training
  Fat and carbohydrate oxidation during exercise measured and estimated with indirect calorimetry.

IPD SHARING:
Plan to Share IPD: No